CLINICAL TRIAL: NCT01515371
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group, 3-stage Dose-finding Study to Identify a Safe and Effective Dose of NT 201 for Unilateral Injection Into the Soft Palate for Treatment of Habitual Snoring
Brief Title: Dose Finding Study for a Botulinum Toxin Type A Injection to Treat Habitual Snoring
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of sufficient eligible subjects, no safety concerns
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201-2069-1; 2011-001779-38 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Habitual Snoring
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IncobotulinumtoxinA (Xeomin) 2.5 Units [U], 5U and 7.4U (Experimental): IncobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kiloDalton), free from complexing proteins") (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection.
  Interventions: Drug: IncobotulinumtoxinA
- Placebo Comparator (Placebo Comparator): Placebo to incobotulinumtoxinA (Xeomin) powder for solution for injection.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Subject to receive one injection of either 2.5U, 5U or 7.4U of IncobotulinumtoxinA.
  For three dose stages: solution prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), reconstitution volume 8 ml, 4 ml and 2.7 ml per 50U vial, respectively, resulting in a concentration of 6.25 U/ml, 12.5 U/ml and 18.5 U/ml. Injection volume is 0.4 ml for all three dose stages. Mode of administration: unilateral soft palate injection.
  Arms: IncobotulinumtoxinA (Xeomin) 2.5 Units [U], 5U and 7.4U
Drug: Placebo Comparator — For three dose stages: solution prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), reconstitution volume 8 ml, 4 ml and 2.7 ml per vial, respectively. Injection volume is 0.4 ml for all three dose stages. Mode of administration: unilateral soft palate injection.
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to identify out of up to three doses a safe and effective dose of Botulinum toxin type A for an injection into one side of the soft palate to treat snoring.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 18-70
* Subjects suffering from snoring for at least 3 months prior to the study start and seeking for help to treat snoring
* Subjects with a peak Snoring Index [SI] ≥ 15/ hour of sleep [h] at baseline visit
* Subjects with a bed partner for at least three months prior to study start.
* Subjects who understand the nature of the study and provide written Informed Consent at screening visit.
* Subjects who understand the study procedures as well as possess the ability and willingness to abide by all procedures during the course of the study

Exclusion Criteria:

* Obese subjects (Body Mass Index ≥ 30)
* Subjects with severe obstructive sleep apnea syndrome
* Subjects with Apnea-Hypopnea Index ≥ 10 /hour of sleep and/ or Respiratory Disturbance Index ≥ 25 / hour of sleep at the baseline visit
* Subjects who have undergone any Botulinum neurotoxin treatment in the history
* Subjects with generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert-Eaton syndrome)
* Acute infections of the pharynx

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in Snoring Index at week 4 | Baseline to week 4
  Snoring Index

SECONDARY OUTCOMES:
Absolute change from baseline in Snoring Index at week 4 | Baseline to week 4
Bed partner satisfaction | Week 4
  Bed partner satisfaction to assess the global effect of the treatment.
Change from baseline in loudness at week 4. | Baseline to week 4
  Sone is employed as the unit of the perceived loudness.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Chair — Merz Pharmaceuticals GmbH
Locations (1):
- Merz Investigational Site #049294, Regensburg, Germany